CLINICAL TRIAL: NCT02481609
Title: Pilot Study of Topical Intranasal N-acetyl Cysteine Administration for the Treatment of Anosmia
Brief Title: NAC Trial for Anosmia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Bradley Goldstein, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130996
Record Dates: First submitted 2015-06-22; First posted 2015-06-25 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Anosmia
Keywords: Loss of Smell; Olfaction; Hyposmia
MeSH Terms: conditions — Anosmia | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NAC arm (Experimental): Topical intranasal N-acetyl cysteine (NAC 200 mg/2 ml vials) BID for one month
  Interventions: Drug: N-acetyl cysteine (NAC)

INTERVENTIONS:
Drug: N-acetyl cysteine (NAC)

SUMMARY:
The purpose of this research study is to evaluate the use of NAC in the treatment of anosmia (a loss of the sense of smell). This drug is already approved by the Food and Drug Administration (FDA) for oral or pulmonary (lung) inhaled use for other medical conditions. However, there is research evidence that the medication may promote nerve recovery (help nerves work better after they are damaged). Since anosmia involves nerve problems, we believe the nasal spray may help treat anosmia. The medication has been in use for many years for other conditions, without safety problems.

ELIGIBILITY:
Inclusion Criteria:

* adults at least 18 years of age with documented microsmia or anosmia by University of Pennsylvania Smell Identification Test.
* patients must have no evidence of active sinonasal disease by nasal endoscopy or CT or MRI
* negative CT or MRI

Exclusion Criteria:

* adults unable to consent
* individuals who are not yet adults (infants, children, teenagers)
* pregnant women, prisoners, employees or subordinates,
* patients with known sensitivity to NAC or severe asthma
* patients with sinus or central disease on CT or MRI imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-07; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Change in the Smell Identification Test score | Baseline and three months after completion of treatment
  Sense of smell is measured using the Smell Identification Test (a standardized 40-item forced choice self administered microencapsulated odor "scratch-and-sniff" style test )

SECONDARY OUTCOMES:
Change in Sino-Nasal Outcome Test (SNOT-20) score | Baseline and three months after completion of treatment
  Validated quality of life assessment tool for nasal and sinus disease patients

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J Goldstein, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miller School of Medicine, Clinical Research Building, Miami, Florida, United States